CLINICAL TRIAL: NCT01557725
Title: Frequency of Vascular Events With Short-term Thromboprophylaxis in Fast-track Hip and Knee-arthroplasty
Acronym: FETA
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Christoffer Joergensen, research fellow/MD, Rigshospitalet, Denmark
Other Study IDs: RH7621
Record Dates: First submitted 2012-03-16; First posted 2012-03-19 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Thromboembolic Events; Post-operative Bleeding
Keywords: Knee Replacement, Total; Hip Replacement, Total; Thromboembolism, Venous; prophylaxis; Enhanced recovery
MeSH Terms: conditions — Thromboembolism; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- THR/TKR patients: Any patients receiving fast-track THR or TKR in departments participating in the Lundbeck Foundation Centre for fast-track THR and TKR

SUMMARY:
There are many different views regarding ideal duration and type of thromboprophylaxis after hip or knee surgery.

An important factor in Fast-track surgery is early mobilization, which in itself is thought to prevent clotting.

The investigators hypothesize that there is no increase with regards to thrombosis in patients receiving fast-track surgery with early mobilization and chemical thrombosis prophylaxis only during hospitalization.

DETAILED DESCRIPTION:
Major orthopaedic surgery is related to development of thrombosis. It is well known that pharmacological prophylaxis reduces the risk of thrombosis after surgery but there are still doubt about the best type of prophylaxis and duration of treatment. The American College of Chest Physicians recommend thromboprophylaxis with either Low molecular weight heparin, factor Xa-inhibitors or Vitamin-K-antagonists for up til 10 days after total knee replacement (TKR) and 35 days after total hip replacement(THR). However whether these recommendations are applicable in fast-track patients receiving early mobilisation is uncertain.

Studies on fast-track patients receiving early mobilisation and thrombosis prophylaxis only during hospitalisation showed very small incidence of symptomatic thromboembolic events. Therefore we conduct a quality-cohort-study on all patients receiving fast-track TKR/THR with short-term anti-thrombotic treatment, in order to investigate frequency of symptomatical deep vein thrombosis, pulmonary embolus, acute myocardial infarction and stroke.

ELIGIBILITY:
Inclusion Criteria:

* primary Uni/bilateral THR/TKR, revision THR/TKR or uni-KR in fast-track setup, Discharged in 3 +-2 days.

Exclusion Criteria:

* not a danish citizen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient receiving elective fast-track THR or TKR
Sampling Method: Non-Probability Sample
Enrollment: 4924 (Actual)
Dates: Start 2010-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Frequency of Vascular events | 90 days postop
  Frequency of symptomatic deep venous thrombosis, pulmonary embolus, acute myocardial infarction, ischemic stroke and other vascular events and/or death

SECONDARY OUTCOMES:
Risk factors of vascular events | 90days postop
  Assessment of preoperative risk factors, and their influence on risk of vascular events after hip and knee arthroplasty

OTHER OUTCOMES:
bleeding events after total hip or knee arthroplasty | 2 days after last dose of prophylaxis
  Assessment of any major bleeding events possibly related to thrombosis prophylaxis after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer C Joergensen, MD, Principal Investigator — Section of surgical pathophysiology, 4074, Rigshospitalet, Copenhagen University, Copenhagen.; Henrik Kehlet, Professor, Study Chair — Section of surgical pathophysiology, 4074 Rigshospitalet, Copenhagen University; Kjeld Soeballe, Professor, Study Chair — Aarhus University hospital, Orthopaedic department E
Locations (6):
- Denmark (6):
  - Aarhus University hospital, Aarhus, Judland
  - Farsoe Hospital, Farsø, Judland
  - Sydvestjydsk Sygehus, Grindsted, Judland
  - Holstebro Hospital, Holstebro, Judland
  - Vejle hospital, Vejle, Judland
  - Hvidovre University hospital, Hvidovre, Region Sjælland

REFERENCES:
- [Background] Petersen PB, Lindberg-Larsen M, Jorgensen CC, Kehlet H; Lundbeck Foundation Centre for Fast-track Hip and Knee Arthroplasty collaborating group. Venous thromboembolism after fast-track elective revision hip and knee arthroplasty - A multicentre cohort study of 2814 unselected consecutive procedures. Thromb Res. 2021 Mar;199:101-105. doi: 10.1016/j.thromres.2021.01.003. Epub 2021 Jan 18. PMID 33485092
- [Background] Petersen PB, Jorgensen CC, Gromov K, Kehlet H; Lundbeck Foundation Centre for Fast-track Hip and Knee Replacement Collaborative Group. Venous thromboembolism after fast-track unicompartmental knee arthroplasty - A prospective multicentre cohort study of 3927 procedures. Thromb Res. 2020 Nov;195:81-86. doi: 10.1016/j.thromres.2020.07.002. Epub 2020 Jul 4. PMID 32673960
- [Background] Petersen PB, Jorgensen CC, Kehlet H; Lundbeck Foundation Centre for Fast-track Hip Knee Replacement Collaborative Group. Venous Thromboembolism despite Ongoing Prophylaxis after Fast-Track Hip and Knee Arthroplasty: A Prospective Multicenter Study of 34,397 Procedures. Thromb Haemost. 2019 Nov;119(11):1877-1885. doi: 10.1055/s-0039-1696686. Epub 2019 Oct 6. PMID 31587249
- [Background] Petersen PB, Kehlet H, Jorgensen CC; Lundbeck Foundation Centre for Fast-track Hip and Knee Replacement Collaborative Group. Safety of In-Hospital Only Thromboprophylaxis after Fast-Track Total Hip and Knee Arthroplasty: A Prospective Follow-Up Study in 17,582 Procedures. Thromb Haemost. 2018 Dec;118(12):2152-2161. doi: 10.1055/s-0038-1675641. Epub 2018 Nov 19. PMID 30453352
- [Background] Jorgensen CC, Kehlet H; Lundbeck Foundation Centre for Fast-track Hip and Knee replacement collaborative group. Early thromboembolic events </=1week after fast-track total hip and knee arthroplasty. Thromb Res. 2016 Feb;138:37-42. doi: 10.1016/j.thromres.2015.12.025. Epub 2015 Dec 29. PMID 26826506
- [Background] Jorgensen CC, Jacobsen MK, Soeballe K, Hansen TB, Husted H, Kjaersgaard-Andersen P, Hansen LT, Laursen MB, Kehlet H. Thromboprophylaxis only during hospitalisation in fast-track hip and knee arthroplasty, a prospective cohort study. BMJ Open. 2013 Dec 10;3(12):e003965. doi: 10.1136/bmjopen-2013-003965. PMID 24334158

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT01557725/Prot_SAP_000.pdf